CLINICAL TRIAL: NCT01435668
Title: Impact Evaluation at 3 Months Follow-up of a Brief Motivational Intervention in Reducing Alcohol Consumption Versus Simple Written Advice Only Among Adolescents Aged 16-24 in Pontchaillou Hospital Emergency Department in Rennes, France
Brief Title: AURAIA Study : Impact Evaluation at 3 Months Follow-up of a Brief Motivational Intervention in Reducing Alcohol Consumption Among Adolescents Aged 16-24 in Pontchaillou Hospital Emergency Department in Rennes, France
Acronym: AURAIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: MAFEJ (Unknown); AIRDDS-CIRDD (Unknown); Observatoire Français des Drogues et des Toxicomanies (OFDT) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LOC/11-01 - AURAIA; 2011-A00017-34 (Other: ID RCB); 11/06-795 (Other: CPP Ouest V (Rennes))
Record Dates: First submitted 2011-09-12; First posted 2011-09-16 (Estimated); Last update posted 2023-03-30 (Actual); Status verified 2014-01

CONDITIONS: Alcohol Abuse, Episodic Drinking Behavior
Keywords: alcohol; hazardous or harmful drinking; emergency department (ED)
MeSH Terms: conditions — Alcoholism; Emergencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Other): A simple written advice.
  Interventions: Behavioral: Simple written advice
- Brief Motivational Intervention (BMI) (Experimental): Brief Motivational Intervention (BMI)
  Interventions: Behavioral: Brief Motivational Intervention (BMI)

INTERVENTIONS:
Behavioral: Brief Motivational Intervention (BMI) — Patients receive an information leaflet plus a referral to a psychologiste. BMI is provided by the psychologist. BMI consists in a first face-to-face interview (35-45 minutes) plus a telephone interview, at 1 and 2 months. Minors' parents are also invited to attend the BMI session.
  Arms: Brief Motivational Intervention (BMI)
Behavioral: Simple written advice — Patients receive an information leaflet.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a Brief Motivational Intervention (BMI), in reducing alcohol consumption among patients with hazardous or harmful drinking admitted in emergency department (ED). Patients aged 16 to 24 and who tested positive for blood alcohol content (BAC) of 0.5g/l. or above are enrolled.

Patients receive either an information leaflet or an information leaflet plus a referral to a psychologist. BMI is provided by the psychologist. BMI consists in a first face-to-face interview (35-45 minutes) plus a telephone interview, at 1 and 2 months. Minors' parents are also invited to attend the BMI session. If necessary, patients can be referred to relevant care and treatment services for alcohol misuse.

In a simple blind, randomised controlled clinical trial of 280 patients, 140 patients are allocated to the treatment group and 140 to the control group. Randomisation is stratified according to patient's age (16-17 or 18-24). Opaque and sealed randomized envelops are used for randomisation.

Alcohol consumption is measured by self-report at 3 months. The principal criteria used to assess the reduction of alcohol use at 3 months follow-up is the number of alcoholic drinks in the last week. Other events such as ED readmission, quarrels related to alcohol, drinking and driving, sexual intercourse without protection will also be assessed. It is the first clinical trial in France comparing these two interventions among young patients in ED with this design.

DETAILED DESCRIPTION:
Eligible patients are recruited by ED physicians. Staff in ED involved in the study is provided with a teaching session on the importance of alcohol misuse and inclusion procedures. Prior to enrolment, a written informed consent is requested from every patient. For patients under 18, a consent form is also requested from parent(s) or the legal tutor.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 16-24 attending ED services between Thursday 10 pm and Sunday 8 am
* Breathalyzer test with a blood alcohol content (BAC) of 0.5g/l or above
* Ability to give consent
* Parental or legal tutor's consent is requested for patients under 18

Exclusion Criteria:

* Already enrolled in the study
* Current ED visit for attempted suicide patients
* Current ED visit for injured trauma patients
* Alcohol dependence requiring hospitalisation or referral to local treatment
* Current enrolment or request to enrol in substance abuse treatment program

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 258 (Actual)
Dates: Start 2011-09; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
alcohol use | 3 months
  The principal criteria used to assess the reduction of alcohol use at 3 months follow-up is the number of alcoholic drinks in the last week. Others indicators such as binge drinking episodes and number of days drinking per week will also be assessed.

SECONDARY OUTCOMES:
ED readmission | 3 months
  ED readmission
quarrels related to alcohol | 3 months
  quarrels related to alcohol
drinking and driving | 3 months
  drinking and driving
sexual intercourse without protection | 3 months
  sexual intercourse without protection

CONTACTS AND LOCATIONS:
Overall Officials: Abdelhouahab BELLOU, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, Brittany Region, France

REFERENCES:
- [Result] Diaz Gomez C, Ngantcha M, Le Garjean N, Brouard N, Lasbleiz M, Perennes M, Kerdiles FJ, Le Lan C, Moirand R, Bellou A. Effect of a brief motivational intervention in reducing alcohol consumption in the emergency department: a randomized controlled trial. Eur J Emerg Med. 2019 Feb;26(1):59-64. doi: 10.1097/MEJ.0000000000000488. PMID 28704267